CLINICAL TRIAL: NCT02286258
Title: MultiGFR: Equivalency Study of Different Methods of Measuring Glomerular Filtration Rate
Brief Title: Validation of New Markers of Glomerular Filtration Rate: Dota Gadolinium and Calcium EDTA (MultiGFR)
Acronym: MultiGFR
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The study was suspended after a suspected unexpected serious adverse event.
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: P100151
Record Dates: First submitted 2014-10-29; First posted 2014-11-07 (Estimated); Last update posted 2018-05-18 (Actual); Status verified 2018-05

CONDITIONS: Renal Insufficiency, Chronic; Kidney Diseases
Keywords: Inulin; Ca-EDTA; Gd-DOTA; Chronic kidney disease; glomerular filtration rate measurement
MeSH Terms: conditions — Renal Insufficiency, Chronic; Kidney Diseases | interventions — Pentetic Acid; Edetic Acid; gadolinium 1,4,7,10-tetraazacyclododecane-N,N',N'',N'''-tetraacetate; gadoterate meglumine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Inuline - Calcium EDTA (Experimental): Calcium EDTA clearance for GFR measurement is compared to inuline clearance in healthy volunteers and CKD patients (stage 1 to 4).
  Interventions: Drug: Calcium EDTA
- Inuline - Gd-DOTA (Experimental): Gd-DOTA clearance for GFR measurement is compared to inuline clearance in healthy volunteers and CKD patients (stage 1 to 4).
  Interventions: Drug: Gd-DOTA

INTERVENTIONS:
Drug: Calcium EDTA — Calcium EDTA for equilibrium GFR measurement : bolus injection 30 mg/kg, then 10 mg/min perfusion for estimated renal clearance 100 mL /min for 4 hours.
  Calcium EDTA for single injection GFR measurement : bolus injection depending on the estimated GFR
  Other Names: Edetic Acid, Calcium, Sodium Salt; Edetate Disodium Calcium
  Arms: Inuline - Calcium EDTA
Drug: Gd-DOTA — Gd-DOTA for equilibrium GFR measurement : bolus injection 56 ng/kg, then 28 ng/min perfusion for estimated renal clearance 100 mL /min for 4 hours.
  Gd-DOTA for single injection GFR measurement : bolus injection depending on the estimated GFR
  Other Names: gadoterate; dotarem; Dota gadolinium
  Arms: Inuline - Gd-DOTA

SUMMARY:
The purpose of this study is to validate in comparison to a reference method (inuline) two novel non-radioactive biomarkers for glomerular filtration rate (GFR) measurement in chronic-kidney disease (CKD) patients and in healthy volunteers: Calcium-EDTA and Gd-DOTA.

DETAILED DESCRIPTION:
Research on estimation and measurement of renal function has been greatly stimulated by the international concept of chronic kidney disease (CKD) and its classification into stages of severity based on the level of glomerular filtration rate (GFR) (National Kidney Foundation KDOQI and ANAES in 2002, KDIGO conference in 2005), and by the development of recommendations for clinical practice according to this stages. Many efforts have focused on the validation of new formula to estimate GFR from endogenous markers. Nevertheless, the performance of these formula is limited by a large inter individual variability, that requires in many cases the use of GFR measurement using exogenous tracers (extreme anthropometric characteristics, abnormal production of endogenous tracers, potential kidney donors, dose adjustment, nephrotoxicity monitoring…). The use of GFR measurement is burdened by a lack of availability due to methodological, biological and regulatory (for radioactive tracers) constraints. That's why a need exists for new validated tracers that will be more accessible and easier to use. Moreover, there are differences between the measurement techniques: single injection of the tracer or concentration equilibrium obtained by continuous infusion; plasma or urinary clearance.

Two new tracers for GFR measurement are here offered for validation: Gd-DOTA and Calcium-EDTA. Gd-DOTA is a macrocyclic paramagnetic contrast product, which can be measured using an ELISA type immunoassay. Although being widely used in radiology with higher doses than those that will be used for GFR measurement in the multi-GFR study, Gd-DOTA has never been involved in systemic nephrogenic fibrosis cases (ProFinest study). Calcium-EDTA has been used for many years for the chelation of heavy metals. Recently, a colorimetric assay for Calcium-EDTA measurement has been developed. Gd-DOTA and Calcium-EDTA clearance for GFR measurement will be compared to inuline clearance in healthy volunteers (25 for each new tracer) and CKD patients (150 for each new tracer).

ELIGIBILITY:
Patients :

Inclusion Criteria:

* males or females without pregnancy
* age : 18-75
* stable chronic kidney disease stages 1 to 4 (MDRD KDIGO 2005), estimated GFR > 15 mL/min/1.73m²
* clinical GFR measurement indication

Exclusion Criteria:

* kidney transplantation
* allergic
* acute disease leading to acute change in GFR
* heavy metals poisoning (treated or not)
* gadolinium contrast agent in the previous month

Healthy volunteers :

Inclusion criteria

* males, 18-35 years old
* weight : 60-100 kg , BMI 18-27 kg/m²
* estimated GFR > 90 mL/min/1.73 m² (MDRD)
* acute diseases in the previous 7 days

Exclusion criteria :

* uro-nephrological disease (past or present)
* nephrotoxic drug chronic use in the previous 2 months
* allergic
* systemic disease (acute or chronic)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Calcium EDTA and Gd-DOTA clearance for glomerular filtration rate measurement | 1 day
  Calcium EDTA or Gd-DOTA clearance for GFR measurement is compared to inuline clearance in healthy volunteers (n= 25) and in CKD patients (n= 150, stages 1 to 4, 30 patients for each stage) at equilibrium by measuring urinary clearances of inuline and Calcium EDTA or Gd-DOTA continuously co-infused after a loading dose.

SECONDARY OUTCOMES:
Calcium EDTA and Gd-DOTA clearance for glomerular filtration rate measurement in each CKD stage | 1 day
  Calcium EDTA or Gd-DOTA clearance for GFR measurement is compared to inuline clearance in healthy volunteers (n= 25) and in CKD patients (n= 150, stages 1 to 4, 30 patients for each stage) at equilibrium by measuring urinary clearances of inuline and Calcium EDTA or Gd-DOTA continuously co-infused after a loading dose.
Calcium EDTA and Gd-DOTA clearance reproducibility for GFR measurement | 15 days
  Calcium EDTA or Gd-DOTA clearance is measured twice at day 1 and day 15 in healthy volunteers (n= 25) and in CKD patients (n= 25, stages 1 to 4, 5 patients for each stage) at equilibrium by measuring urinary clearances of inuline and Calcium EDTA or Gd-DOTA continuously co-infused after a loading dose.
Calcium EDTA and Gd-DOTA clearance with single injection for GFR measurement | 15 days
  Calcium EDTA or Gd-DOTA clearance is measured twice at day 1 and day 15 in healthy volunteers (n= 25) and in CKD patients (n= 25, stages 1 to 4, 5 patients for each stage) at equilibrium at day 1 by measuring urinary clearances of inuline and Calcium EDTA or Gd-DOTA continuously co-infused after a loading dose and at day 15 with a single loading dose of Calcium EDTA or Gd-DOTA
Volumes of distribution of Calcium EDTA and Gd-DOTA | 1 day
  Calcium EDTA or Gd-DOTA apparent volumes of distribution are compared to inuline apparent volume of distribution in healthy volunteers (n= 25) and in CKD patients (n= 150, stages 1 to 4, 30 patients for each stage).
Number of participants with adverse events as a measure of safety. | 45 days
  Each event following Calcium EDTA or Gd-DOTA infusion will be listed in healthy volunteers (n = 50) and in patients (n = 300).

CONTACTS AND LOCATIONS:
Overall Officials: Marie Courbebaisse, Doctor, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (4):
- France (4):
  - Hopital Europeen Georges Pompidou (centre d'investigations cliniques), Paris
  - Hopital Europeen Georges Pompidou (Service de Nephrologie), Paris
  - Hopital Europeen Georges Pompidou (service de Physiologie et des Radioisotopes), Paris
  - CHU Rangueil (service explorations fonctionnelles physiologiques), Toulouse